CLINICAL TRIAL: NCT00972621
Title: Clinical Evaluation of a New Viscoelastic for Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VSCO-106-DISP
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Results first posted 2012-02-22 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrax II (Experimental): Investigational dispersive viscoelastic
  Interventions: Device: Vitrax II
- Viscoat (Active Comparator): Marketed control dispersive viscoelastic
  Interventions: Device: Viscoat

INTERVENTIONS:
Device: Vitrax II — Viscoelastic administered via one or two vials as determined by cataract surgeon for maintenance of anterior chamber.
  Arms: Vitrax II
Device: Viscoat — Currently marketed viscoelastic administered via one or two vials as determined by cataract surgeon for maintenance of anterior chamber..
  Arms: Viscoat

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a new opthalmic viscoelastic material for the use in cataract surgery. The new viscoelastic will be compared to a currently marketed viscoelastic material.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy eye with no pathology other than the presence of cataract
* Visual potential of 20/40 or better

Exclusion Criteria:

* Taking any medications that affect vision, intraocular pressure or ease of cataract surgery (e.g. flomax, glaucoma medications, etc.)
* Known intraocular pressure increases from steroid treatment
* Low endothelial cell count

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AMO Clinical Research Call Center for Trial Locations, Santa Ana, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the general cataract populations from 11 ophthalmic practices between September 2009 and July 2010.
Pre-assignment Details: Enrolled participants who did not meet the inclusion/exclusion criteria as detailed in the protocol were excluded from the trial prior to assignment to study group. Randomization assigned199 Vitrax II subjects and 201 Viscoat subjects, but a randomization error (Viscoat (control) subject treated with Vitrax II) resulted in 200 subjects per group.
Groups:
- Viscoat: Currently marketed viscoelastic
Period: Overall Study
Arm/Group | Vitrax II | Viscoat
Started | 200 | 200
Completed | 200 | 199 (One subject discontinued due to lens exchange.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Results based on safety population (i.e., the population based on the viscoelastic used). If the randomization scheme had been followed correctly, there would have been 199 Vitrax II subjects and 201 Viscoat subjects, but one subject that should have received Viscoat (control treatment) was treated with Vitrax II, which resulted in 200 per group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitrax II | Viscoat | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 54 | 121
  >=65 years | 133 | 146 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.88) | 70.1 (8.86) | 69.03 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 120 | 247
  Male | 73 | 80 | 153
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 400

OUTCOME MEASURES:

1. Primary Outcome: Percent of Intraocular Pressure Spikes 30 mm Hg or Greater Postoperatively
Description: Cumulative rate of Intraoperative Pressure (IOP) spikes 30 mm Hg (millimeters of mercury) or greater measured postoperatively through three months.
Time Frame: 3 months postoperative
Population: Results based on Intent-to-Treat (ITT) population (i.e., population based on the intended randomization scheme, which specified 199 Vitrax II subjects and 201 Viscoat subjects). Study statistical analysis plan specified reporting IOP spikes ≥ 30 mmHg for ITT population, which differs from the safety population used in the Participant Flow.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Vitrax II: Vitrax II: Investigational Treatment
- Viscoat: Viscoat: Control Treatment
Arm/Group | Vitrax II | Viscoat
Number analyzed (Participants) | 199 | 201
percentage of participants | 10.6 [6.97 to 14.14] | 7.6 [4.49 to 10.63]

2. Secondary Outcome: Postoperative Mean Endothelial Cell Count
Description: mean endothelial cell count (measured by Konan specular microscope) at 3 months
Time Frame: 3 months postoperative
Population: Results based on Intent-to-Treat (ITT) population (i.e., population based on the intended randomization scheme, which specified 199 Vitrax II subjects and 201 Viscoat subjects). Study statistical analysis plan specified reporting mean endothelial cell count for ITT population, which differs from the safety population used in the Participant Flow.
Measure: Mean (Standard Deviation); unit: number of endothelial cells
Arm/Group | Vitrax II | Viscoat
Number analyzed (Participants) | 199 | 201
number of endothelial cells | 2454.3 (28.87) | 2366.3 (33.29)

ADVERSE EVENTS:
Arm/Group | Vitrax II | Viscoat
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 21/200 | 15/200
OTHER ADVERSE EVENTS (reported when occurring in more than 4.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitrax II (N=200) | Viscoat (N=200)
IOP Spike greater than or equal to 30 mm HG (Eye disorders) | 21 (22) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least ninety (90) days prior to any proposed submission for publication or presentation of Study Data or other findings related to the Study, Institution will provide Sponsor with a manuscript of such submission(s) for review, comment, and approval.